CLINICAL TRIAL: NCT01350752
Title: A Cost-effectiveness Analysis of Alternative Strategies for the Deployment of ACTs at the Community Level in Cameroon and Nigeria
Brief Title: Research on the Economics of Artemisinin Combination Therapy (ACTs) for the Treatment of Malaria
Acronym: REACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Yaounde (Other); University of Nigeria, Enugu Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REACT
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2013-10

CONDITIONS: Malaria
Keywords: cost effectiveness; provider knowledge; schools
MeSH Terms: conditions — Malaria | interventions — Therapeutics; Quality of Health Care; Longitudinal Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): In Cameroon: Existing practice (with microscopy widely available)
  In Nigeria: Expected practice (RDTs will be provided with basic instructions)
- Provider Intervention (Active Comparator): Cameroon: Introduce malaria RDTs with basic provider training and job aids on malaria diagnosis and treatment. This involved 1-day training on: 1) Malaria Diagnosis; 2) Rapid Diagnostic Testing; 3) Malaria Treatment. These modules explain that all febrile patients should be tested for malaria; procedures for using an RDT; that confirmed cases of uncomplicated malaria should be treated with an ACT; and test-negative patients should not be given an antimalarial.
  Nigeria: Introduce malaria RDTs with provider training and job aids on malaria diagnosis and treatment. This involved a 2-day training workshop and support visits. The training covered the following topics: causes and symptoms of malaria; demonstration on how to use an RDT; updated malaria guidelines; and communications skills. The training used a combination of seminars and facilitated small-group work, such as a treatment algorithm game, problem-solving exercises, self-developed participatory drama and role-playing.
  Interventions: Behavioral: RDTs & Provider Training on Malaria Diagnosis and Treatment
- Extended intervention (Active Comparator): Cameroon: Introduce malaria RDTs with basic provider training and job aids on malaria diagnosis and treatment AND enhanced provider training on improving quality of care. Clinicians received 3-days of training: the first day was identical to the basic intervention, while the remainder of the course covered three additional modules targeting improvements in quality of care: 4) Adapting to Change; 5) Professionalism; 6) Communicating Effectively.
  Nigeria: Introduce malaria RDTs with provider training and job aids on malaria diagnosis and treatment AND School-based malaria education intervention (with drama, peer-health education and distribution of health education materials). In addition, teachers and Peer Health Educators were offered support to hold malaria events in which parents, guardians, and other community members could participate in the same types of activities.
  Interventions: Behavioral: RDTs & Provider Training on Malaria Diagnosis and Treatment; Behavioral: Extended provider training (Cameroon only); Behavioral: School based malaria education (Nigeria only)

INTERVENTIONS:
Behavioral: RDTs & Provider Training on Malaria Diagnosis and Treatment — In Cameroon and Nigeria, malaria RDTs will be made available in health facilities and health care providers will receive training and job aids on malaria diagnosis and treatment. The training course covers the following topics: clinical and parasitological diagnosis of malaria, how to use a rapid diagnostic test, algorithm based on malaria test result, recommended treatment for confirmed malaria cases (including dosage and regimen for artemisinin-based combination therapies), advice for treatment of test-negative patients
  Other Names: RDTs supplied: SD Bioline; Training course
  Arms: Extended intervention; Provider Intervention
Behavioral: Extended provider training (Cameroon only) — 2-day training course which supplements basic provider training on malaria diagnosis and treatment, which focuses on understanding change in malaria treatment guidelines, professionalism, and communication skills
  Other Names: provider training; quality of care
  Arms: Extended intervention
Behavioral: School based malaria education (Nigeria only) — Schools will be invited to undertake activities to raise awareness about malaria RDTs and treatment among children and community members. The intervention includes training teachers on peer health education, malaria awareness activities and providing support to hold a malaria educational event
  Other Names: school based intervention; teachers; peer health educators
  Arms: Extended intervention

SUMMARY:
The objective of the REACT project is to evaluate the effectiveness and cost-effectiveness implications of interventions designed to improve health worker practice in providing treatment for uncomplicated malaria to febrile patients attending health facilities in Cameroon and Nigeria.

DETAILED DESCRIPTION:
NIGERIA

Two interventions will be evaluated: (i) provider intervention including introducing RDTs with detailed instructions, one-off training, job aides and on-the-site supportive supervisory visits and (ii) combined provider intervention [as under (i)]and community-based intervention (using primary and secondary schools as focal points)including school malaria events with drama, peer-health education, distribution of health education materials. Types of facilities include: public primary health facilities, private pharmacies and private Patent Medicine Dealers (PMDs)in Enugu State. The two sites in Enugu State are: Enugu urban (comprising of Enugu East, Enugu South and Enugu North Local government areas (LGA) and Udi LGA. The impact of the interventions will be evaluated using a 3-arm stratified, cluster randomized trial with a cluster defined as a geographical community and the two study sites as the strata. The three arms of the trial are:

* Intervention - Provider intervention
* Intervention - Provider plus school-based malaria activities
* Control - Expected practice (once RDTs have been introduced)

CAMEROON

Two interventions will be evaluated: (i) the introduction of rapid diagnostic tests (RDTs) with basic provider training on malaria diagnosis and treatment; and (ii) the basic provider training [as under (i)] plus enhanced provider training to improve the quality of care that includes aspects of interactive self awareness, communication modules between health workers and also between health workers and patients. Types of facilities include: public district hospitals, public health centres (including integrated health centres), mission hospitals and mission health centres (including integrated health centres)in Yaoundé and Bamenda Health Districts. A stratified, cluster randomized trial will be used in which health facilities are the cluster and the two study sites are the strata. The three arms of the trial are:

* Intervention - RDTs with basic provider training;
* Intervention - RDTs with basic plus enhanced provider training;
* Control - which represents current practice and neither intervention will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* the patient (or their caregiver) reports that the patient is suffering from a fever or has a history of fever in this illness episode
* the patient is present at the health facility

Exclusion Criteria:

* the patient is pregnant
* the patient is <6 months old
* the patient has signs or symptoms of severe malaria

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6513 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Proportion of febrile patients receiving treatment as recommended in clinical guidelines for uncomplicated malaria | As patients exit the health facility
  Recommended treatment is defined as
  * Febrile patients should be tested for malaria, either using microscopy or using a RDT
  * Artemisinin-based Combination Therapy (ACT) should be provided if the patient has a positive malaria test result
  * No antimalarial should be provided if patient has a negative test result.

SECONDARY OUTCOMES:
Health worker knowledge | Two time points: (i) pre and post training evaluation and (ii) during the provider survey (3 months after implementation of interventions)
  Mean score (and standard deviation) in HW knowledge on malaria diagnosis and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Wiseman, Principal Investigator — London School of Hygiene and Tropical Medicine; Wilfred Mbacham, Principal Investigator — University of Yaounde I; Obinna Onwujekwe, Principal Investigator — University of Nigeria
Locations (3):
- Cameroon (2):
  - Various health facilities, Yaoundé, Central Region
  - Various health facilities, Bamenda, North-West Region
- Various health facilities, Enugu, Enugu State, Nigeria

REFERENCES:
- [Derived] Onwujekwe O, Mangham-Jefferies L, Cundill B, Alexander N, Langham J, Ibe O, Uzochukwu B, Wiseman V. Effectiveness of Provider and Community Interventions to Improve Treatment of Uncomplicated Malaria in Nigeria: A Cluster Randomized Controlled Trial. PLoS One. 2015 Aug 26;10(8):e0133832. doi: 10.1371/journal.pone.0133832. eCollection 2015. PMID 26309023
- [Derived] Mbacham WF, Mangham-Jefferies L, Cundill B, Achonduh OA, Chandler CI, Ambebila JN, Nkwescheu A, Forsah-Achu D, Ndiforchu V, Tchekountouo O, Akindeh-Nji M, Ongolo-Zogo P, Wiseman V. Basic or enhanced clinician training to improve adherence to malaria treatment guidelines: a cluster-randomised trial in two areas of Cameroon. Lancet Glob Health. 2014 Jun;2(6):e346-58. doi: 10.1016/S2214-109X(14)70201-3. Epub 2014 Apr 25. PMID 25103303
- [Derived] Achonduh OA, Mbacham WF, Mangham-Jefferies L, Cundill B, Chandler C, Pamen-Ngako J, Lele AK, Ndong IC, Ndive SN, Ambebila JN, Orang-Ojong BB, Metoh TN, Akindeh-Nji M, Wiseman V. Designing and implementing interventions to change clinicians' practice in the management of uncomplicated malaria: lessons from Cameroon. Malar J. 2014 May 29;13:204. doi: 10.1186/1475-2875-13-204. PMID 24885621
- [Derived] Wiseman V, Ogochukwu E, Emmanuel N, Lindsay J M, Bonnie C, Jane E, Eloka U, Benjamin U, Obinna O. A cost-effectiveness analysis of provider and community interventions to improve the treatment of uncomplicated malaria in Nigeria: study protocol for a randomized controlled trial. Trials. 2012 Jun 9;13:81. doi: 10.1186/1745-6215-13-81. PMID 22682276